CLINICAL TRIAL: NCT00735449
Title: Comparing Efficacy and Safety of Combigan With Timolol Adjunctive to Xalatan in Glaucoma or Ocular Hypertension Subjects
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GMA-COM-07-XTC
Record Dates: First submitted 2008-08-13; First posted 2008-08-15 (Estimated); Results first posted 2011-11-24 (Estimated); Last update posted 2019-04-23 (Actual); Status verified 2019-04

CONDITIONS: Glaucoma; Ocular Hypertension
MeSH Terms: conditions — Glaucoma; Ocular Hypertension | interventions — Brimonidine Tartrate, Timolol Maleate Drug Combination; Timolol; Latanoprost

STUDY DESIGN:
Who Masked: Investigator

ARMS (2):
- Combigan ® (Active Comparator): Combigan® (fixed combination of brimonidine tartrate 0.2% timolol maleate 0.5%) adjunctive to Xalatan® (latanoprost 0.005%)
  Interventions: Drug: Fixed combination of brimonidine tartrate 0.2% timolol maleate 0.5%; Drug: latanoprost 0.005%
- Timolol Maleate 0.5% (Active Comparator): Timolol maleate 0.5% adjunctive to Xalatan® (latanoprost 0.005%)
  Interventions: Drug: timolol maleate 0.5%; Drug: latanoprost 0.005%

INTERVENTIONS:
Drug: Fixed combination of brimonidine tartrate 0.2% timolol maleate 0.5% — 1 drop of fixed combination of brimonidine tartrate 0.2% timolol maleate 0.5% taken approximately 12 hours apart, up to 2 times a day.
  Other Names: Combigan®
  Arms: Combigan ®
Drug: timolol maleate 0.5% — 1 drop of timolol maleate 0.5% taken approximately 12 hours apart, up to 2 times a day.
  Other Names: Timpoptic®; Timoptol®
  Arms: Timolol Maleate 0.5%
Drug: latanoprost 0.005% — 1 drop of latanoprost 0.005% once nightly.
  Other Names: Xalatan®

SUMMARY:
Efficacy and safety evaluation of Combigan with timolol when each is used as adjunctive therapy to Xalatan in subjects with glaucoma or ocular hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Be at least 18 years of age
* Give written informed consent
* Be in good general health as determined by your doctor
* Have a diagnosis of unilateral or bilateral glaucoma or ocular hypertension
* If you are a female of child bearing potential, you must be willing to practice effective contraception for the duration of the study (i.e., abstinence, spermicide, condoms, or birth control pills)
* Understand the study instructions, and be able to follow the study instructions; and
* Be likely to complete the entire study period (12 weeks), including all regularly scheduled study visits

Exclusion Criteria:

* Have any active ocular disease other than glaucoma or ocular hypertension that would interfere with study interpretation
* History of severe renal or hepatic impairment
* Subjects with severe cardiovascular disease should not be enrolled unless their disease is controlled and clearance has been obtained from the subject's primary care physician and/or cardiologist
* Contraindications to beta-adrenoceptor antagonist therapy such as chronic obstructive pulmonary disease, bronchial asthma, sinus bradycardia, second and third degree atrioventricular block, overt cardiac failure and cardiogenic shock or uncontrolled congestive heart failure
* Any systemic disease or clinical evidence of any condition which would make the subject, in the opinion of the investigator, unsuitable for the study or could potentially confound the study results; and
* Concurrent participation or prior participation in any investigational drug or device study within the last 30 days prior to the screening visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Actual)
Dates: Start 2008-07; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (2):
- Newark, New Jersey, United States
- Montreal, Quebec, Canada

REFERENCES:
- [Background] Fechtner RD, Harasymowycz P, Nixon DR, Vold SD, Zaman F, Williams JM, Hollander DA. Twelve-week, randomized, multicenter study comparing a fixed combination of brimonidine-timolol with timolol as therapy adjunctive to latanoprost. Clin Ophthalmol. 2011;5:945-53. doi: 10.2147/OPTH.S19999. Epub 2011 Jul 8. PMID 21792284

RESULTS

PARTICIPANT FLOW:
Groups:
- Combigan®: Combigan® (fixed combination of brimonidine tartrate 0.2% timolol maleate 0.5%)adjunctive to Xalatan® (latanoprost 0.005%)
Period: Overall Study
Arm/Group | Combigan® | Timolol Maleate 0.5%
Started | 102 | 102
Completed | 95 | 96
Not Completed | 7 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Combigan® | Timolol Maleate 0.5% | Total
Number analyzed (Participants) | 102 | 102 | 204
Age, Continuous [Median (Full Range); unit: years] | 64.5 [30.1 to 87.0] | 65.9 [29.8 to 88.9] | 65.4 [29.8 to 88.9]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57 | 45 | 102
  Male | 45 | 57 | 102

OUTCOME MEASURES:

1. Secondary Outcome: Mean Intraocular Pressure (IOP) at 10 AM at Week 6
Description: Mean IOP at 10 AM at week 6. IOP is a measurement of the fluid pressure inside the eye.
Time Frame: Week 6
Population: Per-protocol, which included all patients who started the study (randomized) and had at least one follow-up visit.
Measure: Mean (Standard Deviation); unit: Millimeters of mercury (mmHg)
Arm/Group | Combigan® | Timolol Maleate 0.5%
Number analyzed (Participants) | 98 | 97
Millimeters of mercury (mmHg) | 15.9 (3.10) | 16.7 (2.78)

2. Primary Outcome: Mean Intraocular Pressure (IOP) at 10 AM at Week 12
Description: Mean IOP at 10 AM at week 12. IOP is a measurement of the fluid pressure in the eye.
Time Frame: Week 12
Population: Per-protocol, which included all patients who started the study (randomized) and had at least one follow-up visit and who were assessed for this outcome measure at the Week 12 visit.
Measure: Mean (Standard Deviation); unit: Millimeters of mercury (mmHg)
Arm/Group | Combigan® | Timolol Maleate 0.5%
Number analyzed (Participants) | 94 | 94
Millimeters of mercury (mmHg) | 15.1 (2.59) | 16.9 (2.46)

3. Secondary Outcome: Mean Intraocular Pressure (IOP) at 8 AM at Week 12
Description: Mean IOP at 8 AM at week 12. IOP is a measurement of the fluid pressure inside the eye.
Time Frame: Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Millimeters of mercury (mmHg)
Arm/Group | Combigan® | Timolol Maleate 0.5%
Number analyzed (Participants) | 96 | 94
Millimeters of mercury (mmHg) | 17.0 (2.55) | 17.7 (2.58)

4. Secondary Outcome: Mean Intraocular Pressure (IOP) at 8 AM at Week 6
Description: Mean IOP at 8 AM at week 6. IOP is a measurement of the fluid pressure inside the eye.
Time Frame: Week 6
Population: Per-protocol, which included all patients who started the study (randomized) and had at least one follow-up visit.
Measure: Mean (Standard Deviation); unit: Millimeters of mercury (mmHg)
Arm/Group | Combigan® | Timolol Maleate 0.5%
Number analyzed (Participants) | 98 | 97
Millimeters of mercury (mmHg) | 17.3 (2.87) | 17.8 (3.17)

5. Secondary Outcome: Number of Subjects With Adverse Events
Description: Number of subjects with adverse events, defined as any untoward medical occurrence in a subject, during the study (reported through the week 12 visit).
Time Frame: Week 12
Population: Safety population, which included all patients who started the study (randomized) and were treated.
Measure: Number; unit: Participants
Arm/Group | Combigan® | Timolol Maleate 0.5%
Number analyzed (Participants) | 102 | 102
Participants | 15 | 13

ADVERSE EVENTS:
Arm/Group | Combigan® | Timolol Maleate 0.5%
Serious Adverse Events (participants affected / at risk) | 0/102 | 2/102
Other Adverse Events (participants affected / at risk) | 0/102 | 0/102
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Combigan® (N=102) | Timolol Maleate 0.5% (N=102)
Acute exacerbation of COPD (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bacterial bronchitis (Infections and infestations) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo